CLINICAL TRIAL: NCT01209234
Title: Project CLEAR - Changing Lives by Eradicating Antibiotic Resistance
Acronym: CLEAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Susan Huang, Director of Epidemiology and Infection Prevention, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2010-7710
Record Dates: First submitted 2010-09-23; First posted 2010-09-27 (Estimated); Results first posted 2020-09-17 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Methicillin-resistant Staphylococcus Aureus
Keywords: Methicillin-resistant Staphylococcus aureus; MRSA

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MRSA Decolonization (Active Comparator): Participants in this arm will be instructed to complete a decolonization regimen that will involve a 5-day application of nasal mupirocin, oral CHG rinse, and CHG body wash twice a month.
  Interventions: Drug: MRSA Decolonization
- Education Arm (Active Comparator): Patients randomized to standard education will receive a binder with MRSA educational materials which will include or be based upon CDC guidance for MRSA patients at home. In addition, educational material on hygiene practices to prevent MRSA infection will be provided.
  Interventions: Behavioral: Standard-of-Care Education

INTERVENTIONS:
Behavioral: Standard-of-Care Education — Patients randomized to standard education will receive a binder with MRSA educational materials which will include or be based upon CDC guidance for MRSA patients at home.
  Arms: Education Arm
Drug: MRSA Decolonization — Participants in this arm will be instructed to complete a decolonization regimen that will involve a 5-day application of nasal mupirocin, oral CHG rinse, and CHG body wash twice a month.
  Arms: MRSA Decolonization

SUMMARY:
This randomized controlled trial will compare strategies to reduce the risk of methicillin-resistant Staphylococcus aureus (MRSA) infection and re-hospitalization in MRSA carriers. This trial will provide critical answers about the role of decolonization versus standard-of-care education in preventing MRSA infections in the large group of high risk MRSA-positive patients being discharged from hospitals. Findings could potentially impact best practice for the 1.8 million MRSA carriers who are discharged from US hospitals each year.

DETAILED DESCRIPTION:
This randomized controlled trial will compare strategies to reduce the risk of methicillin-resistant Staphylococcus aureus (MRSA) infection and re-hospitalization in MRSA carriers. This trial will provide critical answers about the role of decolonization versus standard-of-care education in preventing MRSA infections in the large group of high risk MRSA+ patients being discharged from hospitals. Findings could potentially impact best practice for the 1.8 million MRSA carriers who are discharged from US hospitals each year.

Specific Aims:

Methicillin-resistant Staphylococcus aureus (MRSA) is arguably the most important single pathogen in healthcare-associated infection when accounting for virulence, prevalence, diversity of disease spectrum, and propensity for widespread transmission. MRSA infection causes or complicates 300,000 hospitalizations each year [Klein, Smith, Laxminarayan], a number which has doubled in the past five years. An additional 1.5 million hospitalized patients either acquire or already harbor the pathogen without current infection. Altogether, these 1.8 million MRSA inpatient carriers experience a high amount of MRSA invasive disease in the year following discharge. Due to increased delivery of complex medical care at home or other post-hospital settings, more and more patients experience serious healthcare-associated morbidity after hospital discharge.[Huang, Platt; Huang, Hinrichsen, Stulgis et al.] In fact, over 80% of patients admitted for MRSA infection have had prior healthcare exposures and are at high risk for repeated MRSA infection.[Huang, Platt; Huang, Hinrichsen, Stulgis et al.; Klevens, Morrison, Nadle, et al.]

Project CLEAR compares two strategies to reduce infection and re-hospitalization due to MRSA among patients being discharged from hospitals. Our trial will compare a long-term regimen aimed at eradicating MRSA body reservoirs with patient education on general hygiene and self care, which is the current standard of care. Our specific aims are:

* To conduct a randomized controlled trial of serial decolonization versus standard-of-care patient education among MRSA carriers upon hospital discharge to reduce post-discharge MRSA infection and re-hospitalization for one year
* To identify predictors of a) infection or re-hospitalization due to MRSA, and b) successful MRSA decolonization, including patient demographics, comorbidities, medical devices, risk behaviors, socioeconomic status, and colonizing MRSA genotype
* To estimate medical and non-medical costs of MRSA infection among MRSA carriers and evaluate the potential for cost savings associated with decolonization

ELIGIBILITY:
Inclusion Criteria:

* 1) At least 18 years old
* 2) Have had a positive culture (a type of test) for MRSA during recent hospital admission or within the 30 days prior to admission or following discharge
* 3) Able to give consent or have a primary caregiver provide consent
* 4) Able to bathe or shower or have this consistently performed by a willing caregiver

Exclusion Criteria:

* 1) Known allergies to chlorhexidine or mupirocin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2140 (Actual)
Dates: Start 2011-01; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan S Huang, MD, MPH, Principal Investigator — University of California, Irivne - School of Medicine
Locations (24):
- United States (24):
  - Covington Care Center, Aliso Viejo, California
  - West Anaheim Extended Care, Anaheim, California
  - Downey Regional Medical Center, Downey, California
  - Fountain Valley Regional Hospital & Medical Center, Fountain Valley, California
  - Orange Coast Memorial Medical Center, Fountain Valley, California
  - St. Jude Medical Center, Fullerton, California
  - Chapman Care Center, Garden Grove, California
  - Pacific Haven HealthCare Center, Garden Grove, California
  - Regents Point at Windcrest, Irvine, California
  - Saddleback Memorial Medical Center - Laguna Hills, Laguna Hills, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - St. Mary Medical Center, Long Beach, California
  - Mission Hospital, Mission Viejo, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Villa Elena Health Care Center, Norwalk, California
  - UC Irvine Medical Center, Orange, California
  - Saddleback Memorial Medical Center - San Clemente, San Clemente, California
  - Little Company of Mary - San Pedro, San Pedro, California
  - Country Villa Plaza, Santa Ana, California
  - Royale Healthcare, Santa Ana, California
  - Torrance Memorial Medical Center, Torrance, California
  - Providence Little Company of Mary Medical Center, Torrance, California
  - Harbor-UCLA Medical Center, Torrence, California
  - Ventura County Medical Center, Ventura, California

REFERENCES:
- [Background] Klein E, Smith DL, Laxminarayan R. Hospitalizations and deaths caused by methicillin-resistant Staphylococcus aureus, United States, 1999-2005. Emerg Infect Dis. 2007 Dec;13(12):1840-6. doi: 10.3201/eid1312.070629. PMID 18258033
- [Background] Huang SS, Platt R. Risk of methicillin-resistant Staphylococcus aureus infection after previous infection or colonization. Clin Infect Dis. 2003 Feb 1;36(3):281-5. doi: 10.1086/345955. Epub 2003 Jan 17. PMID 12539068
- [Background] Huang SS, Hinrichsen VH, Stulgis L, Miroshnik I, Datta R, Watson K, Platt R. Methicillin-resistant Staphylococcus aureus Infection in the Year Following Detection of Carriage (oral presentation). Society of Healthcare Epidemiology of America Annual Meeting (Chicago, IL), March 18-21, 2006.
- [Background] Klevens RM, Morrison MA, Nadle J, Petit S, Gershman K, Ray S, Harrison LH, Lynfield R, Dumyati G, Townes JM, Craig AS, Zell ER, Fosheim GE, McDougal LK, Carey RB, Fridkin SK; Active Bacterial Core surveillance (ABCs) MRSA Investigators. Invasive methicillin-resistant Staphylococcus aureus infections in the United States. JAMA. 2007 Oct 17;298(15):1763-71. doi: 10.1001/jama.298.15.1763. PMID 17940231
- [Derived] Huang SS, Singh R, McKinnell JA, Park S, Gombosev A, Eells SJ, Gillen DL, Kim D, Rashid S, Macias-Gil R, Bolaris MA, Tjoa T, Cao C, Hong SS, Lequieu J, Cui E, Chang J, He J, Evans K, Peterson E, Simpson G, Robinson P, Choi C, Bailey CC Jr, Leo JD, Amin A, Goldmann D, Jernigan JA, Platt R, Septimus E, Weinstein RA, Hayden MK, Miller LG; Project CLEAR Trial. Decolonization to Reduce Postdischarge Infection Risk among MRSA Carriers. N Engl J Med. 2019 Feb 14;380(7):638-650. doi: 10.1056/NEJMoa1716771. PMID 30763195

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between January 10, 2011 and January 2, 2014, during inpatient admissions in 17 hospitals and 7 nursing homes in Southern California.
Period: Overall Study
Arm/Group | MRSA Decolonization | Education Arm
Started | 1070 | 1070
Completed | 1058 | 1063
Not Completed | 12 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MRSA Decolonization | Education Arm | Total
Number analyzed (Participants) | 1058 | 1063 | 2121
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (17) | 56 (17) | 56 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 493 | 480 | 973
  Male | 565 | 583 | 1148
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 840 | 844 | 1684
  Race: Black | 132 | 124 | 256
  Race: Asian | 47 | 58 | 105
  Race: American Indian | 6 | 6 | 12
  Race: Other | 20 | 21 | 41
  Race: Unknown/Not Reported | 13 | 10 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1058 | 1063 | 2121

OUTCOME MEASURES:

1. Primary Outcome: Time to MRSA Infection
Description: Time in days to MRSA inpatient or outpatient infection (analyzed with the use of unadjusted Cox proportional-hazard models to identify time to infection; the results we are reporting are number of participants who had an infection event at one year post discharge)
Time Frame: 1 year
Population: Outcomes were analyzed according to the as-treated adherence strata (fully adherent, partially adherent, and nonadherent participant-time)
Measure: Count of Participants; unit: Participants
Arm/Group | MRSA Decolonization | Education Arm
Number analyzed (Participants) | 1058 | 1063
Participants
  MRSA Infection defined by CDC Criteria | 67 | 98
  MRSA Infection defined by Clinical Criteria | 68 | 98
Statistical Analysis 1: Comparison: MRSA Decolonization vs Education Arm; Test type: Superiority; p = 0.026, Regression, Cox; Cox Proportional Hazard = 0.7, 95% CI 2-sided [0.52 to 0.96], Standard Error of Mean 0.024 — This is the estimated standard error of the log hazard ratio

2. Secondary Outcome: Time to All-cause Infection (Steering Committee Modified Oct 2011)
Description: Time in days to all-cause infection (analyzed with the use of unadjusted Cox proportional-hazard models to identify time to infection; the results we are reporting are number of participants who had an infection event at one year)
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | MRSA Decolonization | Education Arm
Number analyzed (Participants) | 1058 | 1063
Participants
  All-Cause Infection defined by CDC Criteria | 207 | 252
  All-Cause Infection defined by Clinical Criteria | 246 | 298
Statistical Analysis 1: Comparison: MRSA Decolonization vs Education Arm; Test type: Superiority; p = 0.061, Regression, Cox — Not adjusted for multiple comparisons; Cox Proportional Hazard = 0.84, 95% CI 2-sided [0.70 to 1.01], Standard Error of Mean 0.009 — CDC-defined all-cause infection secondary outcome This is the estimated standard error of the log hazard ratio
Statistical Analysis 2: Comparison: MRSA Decolonization vs Education Arm; Test type: Superiority; p = 0.035, Regression, Cox — Not adjusted for multiple comparisons; Cox Proportional Hazard = 0.83, 95% CI 2-sided [0.70 to 0.99], Standard Error of Mean 0.008 — Clinical criteria for all-cause infection This is the estimated standard error of the log hazard ratio

3. Other Pre Specified Outcome: Number of MRSA Infections
Description: Event count of outpatient and inpatient MRSA infections occurring after enrollment
Time Frame: 1 year
Measure: Number; unit: MRSA Infection Events
Arm/Group | MRSA Decolonization | Education Arm
Number analyzed (Participants) | 1058 | 1063
MRSA Infection Events | 67 | 98

4. Other Pre Specified Outcome: Rehospitalization Due to MRSA Infection
Description: Number of participants experiencing rehospitalization due to MRSA infection (first only)
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | MRSA Decolonization | Education Arm
Number analyzed (Participants) | 1058 | 1063
Participants | 57 | 83

5. Other Pre Specified Outcome: Cost and Cost Savings Associated With Post-discharge MRSA Decolonization
Description: Medical and non-medical costs of MRSA infection within the 1 year follow up period
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2027-04

6. Other Pre Specified Outcome: Number of All-cause Infections
Description: Event count of all-cause infections occurring after enrollment
Time Frame: 1 year
Measure: Number; unit: All-cause infection events
Arm/Group | MRSA Decolonization | Education Arm
Number analyzed (Participants) | 1058 | 1063
All-cause infection events | 207 | 252

ADVERSE EVENTS:
Time Frame: Adverse events were actively assessed from January 2011-January 2015. Participants were recruited from January 2011-January 2014 and were followed for 1 year. Evaluation of the full text medical record reviews for adverse events occurred for several years after recruitment ended in 2014.
Arm/Group | MRSA Decolonization | Education Arm
All-Cause Mortality (participants affected / at risk) | 0/1058 | 0/1063
Serious Adverse Events (participants affected / at risk) | 0/1058 | 0/1063
Other Adverse Events (participants affected / at risk) | 48/1058 | 0/1063
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MRSA Decolonization (N=1058) | Education Arm (N=1063)
Nasal Mupirocin (2%) (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) — Congestion
Nasal Mupirocin (2%) (General disorders) | 1 (1) | 0 (0) — Headache
Nasal Mupirocin (2%) (General disorders) | 1 (1) | 0 (0) — Dizziness
Nasal Mupirocin (2%) (General disorders) | 1 (1) | 0 (0) — Numb throat, tast change
Nasal Mupirocin (2%) (General disorders) | 1 (1) | 0 (0) — Runny, itchy nose
Nasal Mupirocin (2%) (General disorders) | 2 (2) | 0 (0) — Runny nose
Nasal Mupirocin (2%) (General disorders) | 1 (1) | 0 (0) — Loss of smell and taste
Chlorhexidine Mouthwash (0.12%) (General disorders) | 1 (1) | 0 (0) — Tongue discoloration
Chlorhexidine Mouthwash (0.12%) (General disorders) | 1 (1) | 0 (0) — Tingling tongue
Chlorhexidine Mouthwash (0.12%) (General disorders) | 1 (1) | 0 (0) — Tingling of mouth
Chlorhexidine Mouthwash (0.12%) (General disorders) | 6 (6) | 0 (0) — Teeth staining
Chlorhexidine Mouthwash (0.12%) (General disorders) | 1 (1) | 0 (0) — Dry mouth
Chlorhexidine Mouthwash (0.12%) (General disorders) | 2 (2) | 0 (0) — Oral irritation
Chlorhexidine Bodywash (4%) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Itchy, dry hands
Chlorhexidine Bodywash (4%) (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — Itchy body
Chlorhexidine Bodywash (4%) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Itchy face and neck
Chlorhexidine Bodywash (4%) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Itchy, dry scalp
Chlorhexidine Bodywash (4%) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Dry skin
Chlorhexidine Bodywash (4%) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Dry, flaky hands and feet
Chlorhexidine Bodywash (4%) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Burning sensation
Chlorhexidine Bodywash (4%) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rash: trunk
Chlorhexidine Bodywash (4%) (Skin and subcutaneous tissue disorders) | 8 (8) | 0 (0) — Rash: body
Chlorhexidine Bodywash (4%) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rash: face and neck
Chlorhexidine Bodywash (4%) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rash: chest
Chlorhexidine Bodywash (4%) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rash: legs
Chlorhexidine Bodywash (4%) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rash: scrotal
Chlorhexidine Bodywash (4%) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rash: neck, limbs
Chlorhexidine Bodywash (4%) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rash and dryness
Chlorhexidine Bodywash (4%) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rash: leg

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2011-04-07): https://cdn.clinicaltrials.gov/large-docs/34/NCT01209234/Prot_000.pdf
  • Statistical Analysis Plan (2012-09-18): https://cdn.clinicaltrials.gov/large-docs/34/NCT01209234/SAP_001.pdf